CLINICAL TRIAL: NCT03163199
Title: TRanslesIonal Assessment of Gradients During Endovascular Therapy
Acronym: TRIAGE
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: CTMS 14-0147-001
Record Dates: First submitted 2017-04-11; First posted 2017-05-22 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Arterial Disease; Fractional Flow Reserve; Hemodynamics
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Translesional Hemodynamic Measurement — Measurement of hemodynamics using the NAVVUS catheter during endovascular therapy

SUMMARY:
Primary objective: To document change in translesional pressure gradients (TLPGs) and ratios (fractional flow reserve) using the NAVVUS RXi catheter following endovascular treatment for symptomatic lower extremity peripheral arterial disease.

Secondary objectives:

* Evaluation of correlation of the ABI and TBI and TLPGs at baseline and following endovascular therapy
* Evaluation of the correlation between the change in WIQ, TCOMs, wound size and change in TLPGS
* Evaluation of correlation between lesion severity by QVA (MLD, % diameter stenosis) and TLPGs
* Evaluation of baseline MLA, MLD, plaque burden by intravascular ultrasound (optional) and TLPGs

DETAILED DESCRIPTION:
There are a lack of tools available for the intraprocedural assessment of endovascular procedures for lower extremity peripheral arterial disease. The present study will use the NAVVUS RXi catheter to document changes in translesional hemodynamics obtained with and without hyperemia in patients undergoing directional atherectomy, angioplasty, and/or stenting of femoropopliteal and infrapoplieal lesions.

ELIGIBILITY:
Inclusions:

* Age >18 y/o, undergoing clinically indicated endovascular therapy (balloon angioplasty, stenting, atherectomy or combination) for lower extremity peripheral artery disease (PAD) and claudication or critical limb ischemia (CLI). Rutherford Category 2-6.
* Includes iliac lesions, common femoral, superficial femoral artery, popliteal artery and tibial vessels
* A subject can be enrolled more than once (up to a maximum of two total times) for treatment of a staged lesion but must wait at least 6 weeks from the completion of the last study enrollment.

Exclusions:

* No pregnant females
* No vulnerable populations (dementia, prisoners, children)
* Baseline bradycardia (heart rate <50 beats/min) or hypotension (systolic blood pressure <90 mm Hg) will be excluded from receiving adenosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with symptomatic peripheral arterial disease (critical limb ischemia or claudication)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Measurement of Change in translesional pressure gradients to determine change in bloodflow with sequential endovascular procedures | At baseline before catheter insertion, after the catheter is first inserted, to obtain initial blood flow reading, then immediately after the each attempt to clear the blockage, up to 5 times during the procedure.
  Observational: • During treatment of Lesion a catheter is inserted into the diseased portion of the artery to remove the plaque and improve the blood flow through the artery. This measurement, which may be repeated 5 times during the treatment, to measure the blood flow at a point before and after the section of the artery with the blockage

CONTACTS AND LOCATIONS:
Overall Officials: Anand Prasad, Principal Investigator — UT Health San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No